CLINICAL TRIAL: NCT06669598
Title: ENHANCING PHYSICAL and COGNITIVE EFFICIENCY in ELDERLY INDIVIDUALS AT RISK of DEMENTIA USING WHOLE-BODY ELECTROMYOSTIMULATION
Brief Title: ENHANCING PHYSICAL and COGNITIVE EFFICIENCY in INDIVIDUALS AT RISK of DEMENTIA USING WHOLE-BODY ELECTROMYOSTIMULATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Molise (Other)
Responsible Party: Principal Investigator, Giuseppe Calcagno, Dott. Prof., University of Molise
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11487/2020
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Mild Cognitive Impairment
Keywords: WB-Electromyostimulation; EMS; electrical muscle stimulation; muscle strength; neurodegenerative disease; cardiovascular training
MeSH Terms: conditions — Cognitive Dysfunction; Neurodegenerative Diseases | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Training Group (Experimental): The ETG group underwent in two 20-minute training sessions per week, with 72 hours of rest between sessions. Each session included aerobic activities such as rowing and treadmill exercises, combined with supervised WB-EMS stimulation. This stimulation utilised a rectangular waveform at 35 Hz, 350 μs, with continuous pulse duration. The intensity of this training modality was set based on heart rate reserve (HRR), starting at 60% HRR in the first week and increasing by 5% every 3 weeks, reaching 80% HRR by the twelfth week.
  Interventions: Other: Whole Body Electromyostimulation
- Control group (Active Comparator): The CON group underwent three weekly training sessions for twelve weeks, con-sisting of 20 minutes of aerobic activity, performed on a treadmill and rowing machine, without the WB-EMS superimposition.
  Interventions: Behavioral: control group

INTERVENTIONS:
Other: Whole Body Electromyostimulation — The ETG group underwent in two 20-minute training sessions per week (12 weeks), with 72 hours of rest between sessions. Each session included aerobic activities such as rowing and treadmill exercises, combined with supervised WB-EMS stimulation. This stimu-lation utilised a rectangular waveform at 35 Hz, 350 μs, with continuous pulse dura-tion
  Arms: Experimental Training Group
Behavioral: control group — The CON group underwent three weekly training sessions for twelve weeks, con-sisting of 20 minutes of aerobic activity, performed on a treadmill and rowing machine, without the WB-EMS superimposition.
  Arms: Control group

SUMMARY:
This study aimed to evaluate the effectiveness of twelve weeks whole-body electrical muscle stimulation combined with aerobic exercises.

DETAILED DESCRIPTION:
This study aimed to evaluate the effectiveness of twelve weeks of WB-EMS (whole-body electrical muscle stimulation at 35Hz and 350 μs) combined with aerobic exercises on a treadmill and rowing machine, in improving physical and cognitive performance in older adults, both healthy and at risk of dementia. The results were compared with those obtained from the same training without WB-EMS.

ELIGIBILITY:
Inclusion Criteria:

* age from 55 to 85 years;
* no simultaneous participation in any type of supervised physical activity;
* Sedentary lifestyle

Exclusion Criteria:

* mini-mental state examination (MMSE) score of less than 24;
* inability to walk for 6 min without assistance;
* the presence of a medical condition influencing the cognitive and/or motor functions;
* the presence of any counter indication for the utilisation of EMS, such as cardiovascular diseases, stents, cardiac pacemakers, and diabetes mellitus, verified by medical certification.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
30-second arm curl test | At the end of 12 weeks
30-second sit-to-stand test | At the end of 12 weeks
hand grip strength test | At the end of 12 weeks
6-minute walking test | At the end of 12 weeks
8-foot up and go test | At the end of 12 weeks
Chair Sit and Reach Test | At the end of 12 weeks
Soda Pop Test | At the end of 12 weeks
Tinetti Balance and Gait Test | At the end of 12 weeks
Mini-Mental State Examination (MMSE) | At the end of 12 weeks
Rey's Auditory Verbal Learning Test (RAVLT) | At the end of 12 weeks
Stroop Colour and Word Interference Test (SCWT) | At the end of 12 weeks
Trail Making Test (TMT) | At the end of 12 weeks
Attentional Matrices Test | At the end of 12 weeks
Prose recall test ( babcock) | At the end of 12 weeks
Frontal Assessment battery (FAB) | At the end of 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi del Molise, Campobasso, CB, Italy

IPD SHARING:
Plan to Share IPD: No